CLINICAL TRIAL: NCT01573507
Title: Neuroprotective Role of Lactate Therapy in Humans With Traumatic Brain Injury
Brief Title: Lactate Therapy After Traumatic Brain Injury
Acronym: LS_TCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Swiss National Science Foundation (Other); European Society of Intensive Care Medicine (Other)
Responsible Party: Principal Investigator, Mauro ODDO, médecin adjoint, PD-MER I, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 237/10
Record Dates: First submitted 2012-04-01; First posted 2012-04-09 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Traumatic Brain Injury; Subarachnoid Hemorrhage
Keywords: traumatic brain injury; lactate; brain metabolism; cerebral microdialysis; subarachnoid hemorrhage; transcranial doppler
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage

STUDY DESIGN:
Intervention Model Description: Hypertonic lactate
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sodium lactate infusion (Experimental): Continuous i.v. infusion of Sodium Lactate (2'400 mOsmol/L) over 3 hours
  Interventions: Other: sodium lactate infusion

INTERVENTIONS:
Other: sodium lactate infusion — 3-6 hours continuous infusion of sodium lactate (20-40 mcg/kg/min)

SUMMARY:
Background: Although glucose is essential to cerebral function, abundant experimental and clinical evidence demonstrates that endogenously released lactate, rather than glucose, is the preferential energy substrate for the brain in conditions of stress and acute injury. In patients with severe Traumatic Brain Injury (TBI) and aneurysmal subarachnoid hemorrhage (SAH) monitored with cerebral microdialysis and brain tissue oxygen (PbtO2), our preliminary data show that increased brain extracellular lactate is frequently observed. Our findings indicate that elevated brain lactate more often occurs in the absence of brain hypoxia/ischemia and is mainly the consequence of increased cerebral glycolysis, i.e. it occurs in association with high extracellular pyruvate. These data suggest that the primary source of elevated lactate is activated glycolysis and strongly support the concept that endogenously released lactate can be utilized by the injured human brain as energy substrate. They prompt further investigation to examine whether exogenous lactate supplementation can be a valuable neuroprotective strategy after TBI or SAH. Indeed, in animal models of brain injury, administration of exogenous lactate improves neuronal and cognitive recovery.

Hypothesis: The investigators test the hypothesis that lactate therapy, administered during the acute phase of TBI or SAH, might exercise neuroprotective actions by restoring brain energetics and improving brain tissue PO2 and cerebral blood flow (CBF).

Aim of the study: The aim of this single-center study is to examine the effect of sodium lactate infusion on cerebral extracellular metabolites, brain tissue PO2 and cerebral blood flow, measured with CT perfusion and transcranial doppler (TCD).

Design: Prospective phase II interventional study examining the effect of a continuous 3-6 hours infusion of sodium lactate (20-40 µmol/kg/min), administered within 48 hours from TBI or SAH, on cerebral extracellular glucose, pyruvate, glutamate, glycerol, PbtO2 and CBF.

DETAILED DESCRIPTION:
Study: Prospective, single-centre phase II interventional study. The study will take place at the Department of Intensive Care Medicine, Lausanne University Medical Center (Centre Hospitalier Universitaire Vaudois, CHUV), Lausanne, Switzerland.

Patient population:

Patients will be monitored with an intra-parenchymal monitoring system, consisting of ICP (Codman®, Integra Neurosciences), PbtO2 (Licox®, Integra Neurosciences) and cerebral microdialysis (CMA Microdialysis®) catheters, based on the protocol for management of TBI presently in use at our center.

Each patient will receive a continuous infusion of sodium lactate (composition: lactate 1'000 mmol/L, Na 1'000 mmol/L: concentration 20-40 µmol/kg/min) for 3-6 hours. Sodium lactate will be prepared locally by the Pharmacie Centrale, CHUV, Lausanne.

Each patient will serve as his/her internal control, and the effect of sodium lactate on all brain physiological variables measured will be anayzed before, during and at the end of sodium lactate infusion.

The main parameters of efficacy are increases of MD glucose, MD pyruvate, PbtO2, and CBF, during sodium lactate perfusion.

For both MD glucose and MD pyruvate, we fixed as the minimal detectable effect of sodium lactate infusion a 30% increase of glucose and pyruvate at the end of the study. To obtain a power of 0.8 with an alpha of 0.05, the number of patients required to complete the study is 33. We therefore plan to include 35 patients.

Statistical analysis: At each time-point (baseline, during perfusion, end of sodium lactate infusion), differences of mean MD glucose, lactate, pyruvate, PbtO2, CBF, Mean transit time, ICP, CPP will be analyzed. We will also examine the percentage time spent with abnormal values (MD glucose < 1 mmol/L, PbtO2 < 20 mm Hg, ICP > 20 mm Hg). Differences will be compared using ANOVA for repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to our intensive care unit (ICU) after severe TBI or poor-grade aneurysmal subarachnoid hemorrhage (SAH), defined by a post-resuscitation Glasgow Coma Scale (GCS) < 9
* Age 18-75 years
* Abnormal head CT-scan (Marshall grade ≥ 2 or Fisher >2)
* Intracranial pressure (ICP), PbtO2 and cerebral MD monitoring as part of standard care

Exclusion Criteria:

* Penetrating TBI
* non aneurysmal SAH
* Age < 18 or > 75 years,
* More than 1 extra-cranial injury with sustained hemodynamic instability and sustained blood lactate elevation > 4 mmol/L
* Cognitive handicap due to previous neurological or neurosurgical history
* Non-survivable injury, brain death or expected death within 48 hours
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Increase from baseline in brain extracellular lactate, pyruvate and glucose | 6 hours
  Increase from baseline in brain extracellular lactate, pyruvate and glucose measured with intra-parenchymal cerebral microdialysis catheter

SECONDARY OUTCOMES:
Increase from baseline in brain tissue PO2 | 6 hours
  Brain tissue PO2 will be measured with intra-parenchymal probes
Increase from baseline in cerebral perfusion pressure | 6 hours
Decrease from baseline in intracranial pressure | 6 hours
plasma sodium | 6 hours
plasma osmolality | 6 hours
mean CBF, measured by transcranial doppler | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Oddo, MD, Principal Investigator — CHUV, Lausanne University Hospital, Switzerland
Locations (1):
- CHUV, Lausanne University Hospital, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carteron L, Solari D, Patet C, Quintard H, Miroz JP, Bloch J, Daniel RT, Hirt L, Eckert P, Magistretti PJ, Oddo M. Hypertonic Lactate to Improve Cerebral Perfusion and Glucose Availability After Acute Brain Injury. Crit Care Med. 2018 Oct;46(10):1649-1655. doi: 10.1097/CCM.0000000000003274. PMID 29923931
- [Derived] Bouzat P, Sala N, Suys T, Zerlauth JB, Marques-Vidal P, Feihl F, Bloch J, Messerer M, Levivier M, Meuli R, Magistretti PJ, Oddo M. Cerebral metabolic effects of exogenous lactate supplementation on the injured human brain. Intensive Care Med. 2014 Mar;40(3):412-21. doi: 10.1007/s00134-013-3203-6. Epub 2014 Jan 30. PMID 24477453